CLINICAL TRIAL: NCT05319327
Title: Targeting DNA-methylation Fingerprints Linked to Ultra-Processed Foods Consumption to Prevent Non-communicable Diseases: the METHYL-UP Study
Acronym: METHYL-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Responsible Party: Principal Investigator, Lidia Daimiel Ruiz, Senior Researcher, IMDEA Food
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMD: PI-048
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Overweight
Keywords: Epigenetics; Methylation; Clinical trial; Causal inference; Non-communicable diseases; Precision nutrition; Ultra-processed food; NOVA; Obesity
MeSH Terms: conditions — Obesity; Overweight; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, parallel groups intervention
Who Masked: Investigator
Masking Description: The investigator who will analyze data will be provided with blinded data regarding the groups. Control and intervention groups will be randomly designated as group A and B. Investigator responsible for the analyses of the effect of the intervention on primary outcomes will compared groups A and B in a blinded manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group will be provided with nutritional guidelines to follow a healthy diet based on a Mediterranean diet.
  Interventions: Other: Control
- Intervention group (Experimental): Participants in the intervention group will follow a nutritional intervention program aimed to reduce UPF consumption. Nutritional intervention will not modify basal caloric intake but will record energy intake along the intervention. Nutritional counseling will be based on nutritional educational material such as encouraged and discouraged food items, recipes, menus and food shopping lists based on unprocessed or minimally processed foods.
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — A nutritional intervention program aimed to reduce UPF consumption. Nutritional intervention will not modify basal caloric intake but will record energy intake along the intervention. Nutritional counseling will be based on nutritional educational material such as encouraged and discouraged food items, recipes, menus and food shopping lists based on unprocessed or minimally processed foods.
  Total intervention will last 6 months for both groups. During the intervention phase, a monthly interview with nutritionist/dietitian is scheduled. Face-to-face interviews will be carried out in months 2 and 4. Phone interviews will be carried out in months 1, 3 and 5. In the baseline and final visits (months 0 and 6) a sample and data collection will be performed.
  Other Names: Reduction of UPF consumption
  Arms: Intervention group
Other: Control — General counseling to adhere to a healthy Mediterranean diet
  Arms: Control Group

SUMMARY:
Non-communicable diseases (NCD) are the main health challenge in industrialized countries. However, these diseases are preventable if an intervention based on lifestyle is implemented at the population level. Diet has a great impact on the onset and progression of NCD. In this regard, ultra-processed food (UPF) consumption has been related to higher morbidity and mortality. UPF are defined as "formulations made mostly or entirely from substances derived from foods and additives, with little if any intact unprocessed or minimally processed foods" (NOVA definition). UPF are rich in saturated fats and additives and poor in fiber other nutrients. UPF consumption has raised in the last decades in the industrialized countries and this increase has been associated with higher prevalence of metabolic disorders such as diabetes, obesity, metabolic syndrome, cardiovascular disease, and cancer. However, mechanisms that link UPF consumption with NCD are poorly understood and clinical trials are needed to unravel these mechanisms and how to impact on them through lifestyle interventions. The investigators have previously identified DNA methylation marks associated with UPF consumption. DNA methylation marks are modifiable. The aim of the study is to assay if DNA methylation marks related to UPF consumption are reversible by reducing UPF consumption in a population of adults with overweight or obesity and with a high basal UPF consumption (>35% of total food consumption in g/day).

DETAILED DESCRIPTION:
The investigators propose a controlled, randomized, parallel groups intervention study based on nutritional counseling to reduce UPF consumption. Eligible participants are adults (18-50 years old), men and women, with overweight or obesity (BMI 25-40 Kg/m2) with a high basal consumption of UPF (>35% of total intake in g/day).

Recruited participants will be randomly allocated into a control group or an intervention group. Participants in the control group will be provided with nutritional guidelines to follow a healthy diet based on a Mediterranean diet. Participants in the intervention group will follow a nutritional intervention program aimed to reduce UPF consumption. Nutritional intervention will not modify basal caloric intake but will record energy intake along the intervention. Nutritional counseling will be based on nutritional educational material such as encourage and discourage food items, recipes, menus and food shopping lists based on unprocessed or minimally processed foods.

Total intervention will last 6 months for both groups. During the intervention phase, a monthly interview with nutritionist/dietitian is scheduled. Face-to-face interviews will be carried out in months 2 and 4. Phone interviews will be carried out in months 1, 3 and 5. In the baseline and final visits (months 0 and 6) a sample and data collection will be performed.

Data collected will include general socio-demographical data (age, sex, educational level, working status, civil status, rural/urban status), lifestyle data (smoking habits, dietary habits, physical activity, sleeping habits), anthropometric data (height, weight, waist circumference, body composition), and clinic-phenotypical parameters (blood pressure, medication, adverse effects, disease prevalence). Biological sample collection will include blood, urine, saliva and feces. Biochemical and blood cells parameters will be measured (blood cell count, glucose, lipid and hepatic profiles).

ELIGIBILITY:
Inclusion Criteria:

* Men/women
* 18-50 years old
* BMI 25-40 Kg/m2
* UPF consumption > 35% of total intake in g/day

Exclusion Criteria:

* Pregnancy
* Menopause
* IMC <25 Kg/m2 or > 40 Kg/m2
* Excessive alcohol consumption
* Prevalent cardiovascular, renal, lung, pancreatic or liver disease
* Type 1 diabetes
* Type 2 diabetes with poor glucose control or unstable medication during last 3 months
* Prevalent endocrine disease
* Changes in anti-hypertensive medication during last 3 months
* Insulin, systemic anti-inflammatory, or glucocorticoid medication during last 3 months
* Food allergies or intolerances
* Psychosocial or cultural factors that prevent from following the intervention

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
UPF | 6 months
  Ultra-processed food consumption

SECONDARY OUTCOMES:
Weight | 6 months
  Weight change (Kg)
BMI | 6 months
  Change in body mass index (Kg/m2)
Obesity | 6 months
  Percentage of participants who reverse obesity condition (BMI < 30 Kg/m2)
Body composition | 6 months
  Change in % of fat mass

OTHER OUTCOMES:
DNA methylation | 12 months
  Reversibility of DNA methylation marks
Glucose | 9 months
  Change in fastin glucose levels (mg/dL)
Glycated haemoglobin | 9 months
  Change in fastin glycated haemoglobin levels (%)
Triglycerides | 9 months
  Change in fasting triglycerides levels (mg/dL)
LDL-cholesterol | 9 months
  Change in fasting LDL-cholesterol levels (mg/dL)
HDL-cholesterol | 9 months
  Change in fasting HDL-cholesterol levels (mg/dL)
Liver profile | 9 months
  Change in HSI liver function index
Microbiota | 24 months
  Changein microbiota diversity

CONTACTS AND LOCATIONS:
Overall Officials: José M Ordovás, PhD, Study Director — Fundación IMDEA Alimentación
Locations (1):
- IMDEA Food, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Informed consent does not allow to make data publicly available. Nevertheless, data could be share upon request to the investigators.

REFERENCES:
- See also: Research team profile — https://www.food.imdea.org/nutritional-genomics-and-epigenomics-group
- See also: Research team profile — https://www.food.imdea.org/nutritional-control-epignome